CLINICAL TRIAL: NCT05991089
Title: Tunisian Clinical Registry on Chronic Kidney Disease in Hypertensive Patients. National Multicentric Cross Section Survey.
Brief Title: Tunisian Clinical Registry on Chronic Kidney Disease in Hypertensive Patients
Acronym: TUN-CKDH
Status: Completed | Type: Observational
Sponsor: Dacima Consulting (Other)
Collaborators: Tunisian Society for Nephrology, Dialysis and Renal Transplantation (Unknown)
Responsible Party: Sponsor
Other Study IDs: DAC-014-TUNCKDH
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases; Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In Tunisia, high blood pressure (HTN) is a public health problem whose prevalence varies from 28.7% to 34.7%. Hypertension can be both, cause and consequence of chronic kidney disease, and its prevalence is quite high in this population. It is both a risk factor for mortality and cardiovascular morbidity, but also a major cause of terminal chronic kidney disease becoming an additional public health concern.

Detecting and diagnosing chronic kidney in all hypertensives at an early stage remains a global public health challenge. A well-conducted treatment makes it possible to reach the blood pressure objective but also to reduce the risk of occurrence of a cardiovascular event and to slow the progression of chronic kidney disease.

In Tunisia, few data exists concerning the prevalence of chronic kidney disease in hypertensive subjects, thus limiting the development and elaboration of preventive measures. A national survey will thus be conducted by the "Kidney and Metabolic Diseases" Working Group under the aegis of the Tunisian Society of Nephrology, Dialysis and Kidney Transplantation. The main objective is to estimate the prevalence of chronic kidney disease in hypertensive tunisian patients.

DETAILED DESCRIPTION:
This is national multicentric cross-sectional survey. The study will be carried out for one month at medical departments and ambulatory clinics of general physicians, family medicine specialists, endocrinologists, specialists in nutrition and metabolic diseases, nephrologists, internal medicine physicians, cardiologists, all physicians caring for non-diabetic hypertensive patients or any healthcare providers in charge of hypertensive patients.

A Steering Committee helps investigators to monitor their patient inclusions, performs audit trails and prepares the statistical analysis plan for the study. Collected data are managed by the DACIMA Clinical Suite®, the electronic data capture platform which complies with the FDA 21 CFR part 11 requirements (Food and Drug Administration 21 Code of Federal Regulations part 11), the HIPAA specifications (Health Insurance Portability and Accountability Act), and the ICH standards (International Conference on Harmonisation).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Hypertension
* Follow-up at consultation at least for three months before enrollment date
* Informed consent

Exclusion Criteria:

* Hypertension emergency
* Pregnancy
* Kidney transplanted subjects
* Dialysis stage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All confirmed hypertensive patients at enrollment
Sampling Method: Non-Probability Sample
Enrollment: 11770 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of Chronic Kidney Disease | At inclusion
  Frequency of hypertensive subjects with chronic kidney disease

CONTACTS AND LOCATIONS:
Overall Officials: Jannet Labidi, MD, Study Chair — Military Hospital of Tunis (Tunis, Tunisia); Amel Harzallah, MD, Principal Investigator — University Hospital of Charles Nicolle (Tunis, Tunisia); Awatef Azzabi, MD, Principal Investigator — University Hospital of Sahloul (Sousse, Tunisia); Badreddine Ben Kaab, MD, Principal Investigator — La Marsa Internal Security Forces Hospital (Tunis, Tunisia); Ikram Mami, MD, Principal Investigator — University Hospital of La Rabta (Tunis, Tunisia); Lamia Rais, MD, Principal Investigator — University Hospital of La Rabta (Tunis, Tunisia); Maissa Hadji Brahim, MD, Principal Investigator — University Hospital of Taher Sfar (Mahdia, Tunisia); Mouna Hammouda, MD, Principal Investigator — University Hospital of Fattouma Bourguiba (Monastir, Tunisia); Sahar Agrebi, MD, Principal Investigator — University Hospital of Charles Nicolle (Tunis, Tunisia); Seifeddine Azaiez, MD, Principal Investigator — Private Clinic (Ben Arous, Tunisia); Soumaya Chargui, MD, Principal Investigator — University Hospital of Charles Nicolle (Tunis, Tunisia)
Locations (1):
- Tunisian Society for Nephrology, Dialysis and Renal Transplantation, Tunis, Tunisia, Tunisia

IPD SHARING:
Plan to Share IPD: No